CLINICAL TRIAL: NCT00393068
Title: A Phase II Trial of Preoperative Concurrent Chemotherapy/Radiation Therapy Plus Bevacizumab/Erlotinib in the Treatment of Localized Esophageal Cancer
Brief Title: Chemotherapy, Radiation Therapy and Immunotherapy Prior to Surgery in Operable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 91
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab; Paclitaxel; Carboplatin; Fluorouracil; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Prior to surgery study treatment will be given over a 6 weeks (Days 1-42) period. Beginning Day 1 and continuing through Day 35 patients will receive a continuous infusion of 5-FU by vein. A small portable pump will be used to administer this drug into a tube that has been surgically inserted into the patient's vein. On Day 1 and 22 patients will also receive the drugs paclitaxel, carboplatin and bevacizumab by vein. Erlotinib is given by mouth beginning on Day 1 and continuing through Day 45. Patients will receive radiation therapy daily, Monday through Friday, beginning Day 1-35 (approximately 5 weeks).
  Surgery will be performed approximately 12-14 weeks after beginning this combined treatment.
  Interventions: Drug: Erlotinib; Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: 5-FU; Procedure: Radiation therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Erlotinib — Erlotinib
  Other Names: Tarceva
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel
  Other Names: Taxol
Drug: Carboplatin — Carboplatin
  Other Names: Paraplatin
Drug: 5-FU — 5-FU
  Other Names: Fluorouracil
Procedure: Radiation therapy — Radiation therapy
Procedure: Surgery — Surgery

SUMMARY:
The purpose of this study is to see if adding two targeted drugs (bevacizumab and erlotinib) further improves the response to chemotherapy (5-FU, paclitaxel, carboplatin) and radiation therapy in patients with operable esophageal cancer.

Side effects (toxicity) information will also be collected.

DETAILED DESCRIPTION:
Surgical removal has been the standard treatment for operable esophageal cancer. However, recent studies have shown improved results when patients receive a short course of chemotherapy and radiation therapy prior to surgery.

Prior to surgery study treatment will be given over a 6 weeks (Days 1-42) period. Beginning Day 1 and continuing through Day 35 patients will receive a continuous infusion of 5-FU by vein. A small portable pump will be used to administer this drug into a tube that has been surgically inserted into the patient's vein. On Day 1 and 22 patients will also receive the drugs paclitaxel, carboplatin and bevacizumab by vein. Erlotinib is given by mouth beginning on Day 1 and continuing through Day 45. Patients will receive radiation therapy daily, Monday through Friday, beginning Day 1-35 (approximately 5 weeks).

Surgery will be performed approximately 12-14 weeks after beginning this combined treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed esophageal or gastroesophageal junction cancer stage I, II or III
* No prior treatment for esophageal cancer
* Must be surgical candidate based on stage and location of disease
* Measurable or evaluable disease
* Able to be up and perform self care
* Adequate liver, renal function and bone marrow function
* Patients will have to have a central venous access device placed
* Able to give written informed consent.
* Age 18 or older

Exclusion Criteria:

* Stage IV disease
* Prior cancer treatment for advanced cancer in the last 5 years
* Pregnant or lactating women
* History of stroke, transient ischemic attacks, or acute MI within the past 6 months or any other serious cardiovascular disease
* History of neurological disease
* Recent history of blood in the sputum or vomitus
* Non-healing wounds, ulcer or long bone fractures
* History of bleeding problems or coagulation problems
* History of abdominal fistula, gi perforation or intrabdominal abscess within 6 months
* History of uncontrolled hypertension

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Aultman Hospital, Canton, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Bendell JC, Meluch A, Peyton J, Rubin M, Waterhouse D, Webb C, Burris HA 3rd, Hainsworth JD. A phase II trial of preoperative concurrent chemotherapy/radiation therapy plus bevacizumab/erlotinib in the treatment of localized esophageal cancer. Clin Adv Hematol Oncol. 2012 Jul;10(7):430-7. PMID 22895283

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 62
Completed | 44
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 64 [43 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 57
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: pCR was defined as no residual viable cancer found at the primary site or regional lymph nodes upon pathologic review of the surgical specimen for patients who went to surgical resection.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 62
Participants | 18

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time interval from the start of treatment until death. Patients who remained alive were censored at the date of their last tumor assessment.
Time Frame: 32 months
Population: All patients receiving a dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 62
months | 30.16 [19.35 to NA] — Upper confidence limit is not estimable by Kaplan-Meier method due to insufficient observed events.

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from the date of first treatment until the date of disease progression or death, whichever occurred first. Patients who did not progress were censored at the date of their last tumor assessment.
Time Frame: 36 months
Population: All patients receiving a dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 62
months | 28.58 [14.39 to NA] — Upper confidence limit is not estimable by Kaplan Meier method due to insufficient observed events.

ADVERSE EVENTS:
Time Frame: 32 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 29/62
Serious Adverse Events (participants affected / at risk) | 38/62
Other Adverse Events (participants affected / at risk) | 59/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=62)
Leukocytes (Blood and lymphatic system disorders) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 6 (6)
Supraventricular arrhythmia - atrial fibrillation (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Peripheral Arterial Ischemia (Vascular disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 5 (6)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
GI - Other (Gastrointestinal disorders) | 1 (1) — Severe Odynophagia
Malnutrition (Gastrointestinal disorders) | 1 (1)
Hemorrhage - GI (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Adult Respiratory Distress Syndrome
Intraop Injury - Abdominal (Surgical and medical procedures) | 2 (2)
Intraop Injury - Esophagus (Surgical and medical procedures) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=62)
Leukocytes (Blood and lymphatic system disorders) | 40 (40)
Neutrophils (Blood and lymphatic system disorders) | 27 (27)
Platelets (Blood and lymphatic system disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Mucositis - Oral Cavity (Gastrointestinal disorders) | 26 (26)
Dehydration (Gastrointestinal disorders) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Esophagitis (Gastrointestinal disorders) | 17 (17)
Anorexia (Gastrointestinal disorders) | 10 (10)
Fatigue (General disorders) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 4 (4)
Hemorrhage - GI (Gastrointestinal disorders) | 3 (3)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.